CLINICAL TRIAL: NCT01091805
Title: Correlation of Oropharyngeal Pepsin and Gastroesophageal (GE) Reflux
Acronym: Pepsin
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00006309
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2013-03

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to see if GE reflux events are associated with increasing levels of pepsin in spit samples. Pepsin is a special protein called an "enzyme" that is made only in your stomach. It is not normally found in your throat. Pepsin breaks down food proteins that you eat to form nutritional building blocks that your body can use to grow. An enzyme is a substance that helps break down proteins.

Gastroesophageal reflux disease (GERD) is very common in infants and children, but can result in serious health problems if not accurately diagnosed. The investigators currently do not have a definitive test to be used as a standard for diagnosing pediatric GERD.

Measurement of pepsin, an enzyme normally produced only in the stomach, has been used as a non-invasive way to detect gastric aspiration (reflux of stomach fluid into the airway) in both adults and children, but using pepsin to detect reflux has not been tested. Since pepsin should not be present in the normal esophagus and respiratory tract, but is always present in reflux fluid from the stomach, the investigators believe that the more GE reflux the investigators detect, the higher the levels of pepsin the investigators see in the fluid collected from the mouth. If patients do not have GE reflux, but have swallowing problems alone in which food or liquid goes into the airway, the investigators expect that these patients will have no pepsin in the fluid collected from their mouth.

The investigators will test these hypotheses by measuring pepsin levels from mouth fluid and comparing them with the number of GE reflux events the investigators find using the pH/impedance (MII (multichannel intraluminal impedance)) test. Since the investigators are interested in pepsin levels for all types of reflux - acid and non-acid -the investigators will study children whether or not they are on acid blocking medicines. The investigators will also look at pepsin levels in patients whose pH/MII is normal, but have aspiration alone that the investigators find on a modified barium swallow (MBS) study. The investigators will measure pepsin levels in healthy children with no reflux symptoms and no swallowing problems as the investigators controls. The investigators anticipate that this study will show a positive correlation between GE reflux events and the presence of oropharyngeal pepsin, which may allow us to use pepsin as a way to test for reflux.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients from birth to 18 years (including premature infants) who are deemed clinically to require 24 hour esophageal pH/impedance.
2. Pediatric patients (newborn to 18 years) undergoing MBS who have had or will have pH/MII monitoring within 6 months.
3. Patients' parents or legal guardians will provide written informed consent for the protocol. When appropriate, patient assent will be obtained.

Exclusion Criteria:

1. Patients with anatomic facial anomalies or facial discomfort precluding nasal intubation of the pH/MII catheter.
2. Patient unable to complete a 24 hour pH/MII study.
3. Children fed exclusively with nasogastric or nasojejunal (transpyloric) tube at the time of study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Wake Forest University Baptist Medical Center, Section of Gastroenterology Pediatric Clinic
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Positive correlation between GE reflux events and oropharyngeal pepsin concentrations | 24 Hours
  1. Total number of GE reflux events by MII over 24 hours. Events will be further subdivided into acid or non-acid based on distal pH measurements.
  2. Total number of GE reflux events by MII over 24 hours will be classified as distal, mid, or proximal esophagus. Proximal events will be classified as acid or non-acid based on proximal pH sensor recordings.
  3. Esophageal clearance time for all GE reflux events.
  4. Oropharyngeal pepsin concentration immediately before and 30 minutes after feeds.
  5. Oropharyngeal pepsin concentration after awakening.
Compare oropharyngeal pepsin concentrations in patients with GE reflux to a. patients with normal pH/MII and isolated oral aspiration on MBS b. healthy controls. | 24 hours

SECONDARY OUTCOMES:
Non-acid GE reflux events are positively correlated with increasing levels of oropharyngeal pepsin. | 24 hours
  1. Total number of GE reflux events by MII over 24 hours. Events will be further subdivided into acid or non-acid based on distal pH measurements.
  2. Total number of GE reflux events by MII over 24 hours will be classified as distal, mid, or proximal esophagus. Proximal events will be classified as acid or non-acid based on proximal pH sensor recordings.
  3. Esophageal clearance time for all GE reflux events.
  4. Oropharyngeal pepsin concentration immediately before and 30 minutes after feeds.
  5. Oropharyngeal pepsin concentration after awakening.
Patients with isolated oral aspiration (without GE reflux) will have no oropharyngeal pepsin. | 24 hours
  1. Total number of GE reflux events by MII over 24 hours. Events will be further subdivided into acid or non-acid based on distal pH measurements.
  2. Total number of GE reflux events by MII over 24 hours will be classified as distal, mid, or proximal esophagus. Proximal events will be classified as acid or non-acid based on proximal pH sensor recordings.
  3. Esophageal clearance time for all GE reflux events.
  4. Oropharyngeal pepsin concentration immediately before and 30 minutes after feeds.
  5. Oropharyngeal pepsin concentration after awakening.

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Fortunato JE, D'Agostino RB Jr, Lively MO. Pepsin in saliva as a biomarker for oropharyngeal reflux compared with 24-hour esophageal impedance/pH monitoring in pediatric patients. Neurogastroenterol Motil. 2017 Feb;29(2). doi: 10.1111/nmo.12936. Epub 2016 Sep 7. PMID 27604397